CLINICAL TRIAL: NCT04549922
Title: Antisense Therapy to Block the Kallikrein-kinin Pathway in COVID-19: A Phase II Randomized Controlled Trial
Brief Title: Antisense Therapy to Block the Kallikrein-kinin Pathway in COVID-19
Acronym: ASKCOV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry); Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASKCOV_Trial
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: antisense; kallikrein-kinin
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo used in the present study will consist of 0.9% NaCl Solution, which has the same physical characteristics as the ISIS 721744 drug. The placebo solution will be prepared by the nurse or pharmacist of the research team at the time of application. The nurse will be trained on the procedures for adequate blinding of the intervention. The pharmacist at the site level will not be blind, but the rest of the ream (nurse, physicians, patients, etc) will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1.2 mL Normal Saline, single dose subcutaneous, after randomization
  Interventions: Drug: Normal Saline
- ISIS 721744 (Active Comparator): 1.2 mL ISIS 721744, single dose subcutaneous, after randomization
  Interventions: Drug: ISIS 721744

INTERVENTIONS:
Drug: ISIS 721744 — 1.2 mL of ISIS 721744 subcutaneous once after randomization
  Arms: ISIS 721744
Drug: Normal Saline — 1.2 mL subcutaneous
  Arms: Placebo

SUMMARY:
Up to 1/3 of all patients infected with COVID-19 can develop complications that require hospitalization. Severe pneumonia associated with acute respiratory distress syndrome (ARDS) is the most threatening and feared complication of COVID-19 infection, with mortality rates close to 50% in some groups.

Autopsies between these severe cases reveal severe capillary involvement, with signs of intense inflammatory changes, microvascular thrombosis, endothelial injury and abnormal tissue repair. The available evidence suggests that abnormal activation or imbalance in the counter-regulation of the kallikrein-kinin system may play a central role in a positive feedback cycle, leading to consequent diffuse microangiopathy. Blockade of the kallikrein-kinin system can therefore prevent deterioration of lung function by reducing inflammation, edema and microthrombosis.

The objective of this phase IIb study is to assess the preliminary effects on the oxygenation parameters of an antisense oligonucleotide that inhibits pre-kallikrein synthesis in patients with moderate to severe COVID-19.

DETAILED DESCRIPTION:
The objective of this phase IIb study is to assess the preliminary effects on the oxygenation parameters of an antisense oligonucleotide that inhibits pre-kallikrein synthesis in patients with moderate to severe COVID-19.

This is a blind randomized pilot clinical study which aims to include 110 patients (55 per arm).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with COVID-19 who need supplemental oxygen
2. Women must not be pregnant or breastfeeding, and must be surgically sterile or in the postmenopausal stage (without risk of becoming pregnant).
3. Men must be surgically sterile or abstinent or, if they are having sex with risk of pregnancy, the subject must use an effective method of contraception from the moment they sign the informed consent form until at least 24 weeks after the dose of the study drug (ISIS 721744 or placebo).

Exclusion Criteria:

1. Patients on invasive mechanical ventilation or who may need mechanical ventilation for the next 24 hours. The use of non-invasive ventilation and/or a high-flow nasal catheter is permitted.
2. Patients with > 10 days since symptom onset or more than 48h of oxygen use
3. Pregnancy, breast-feeding or risk of becoming pregnant
4. Hemodynamically unstable (use of vasoconstrictors, such as norepinephrine, at any dose)
5. Previous diagnosis of heart failure at functional class III or IV
6. Previous uncontrolled hypertension (more than 3 drug classes use at home)
7. Severe lung disease (use of home oxygen)
8. Age < 18 and > 80 years
9. Physician and family not committed to full life support and/or with severe existing illness with a life expectancy of less than 12 months
10. Refusal to accept informed consent and/or unwillingness to comply with all requirements of the study procedure and security monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Days alive without respiratory support (any supplemental oxygen) after 15 days (DAFOR15) | 15 days
  Number of days the patient is alive and not receiving any supplementary respiratory support (oxygen, non-invasive ventilation, high flow nasal catheter or mechanical ventilation) during 15 days

SECONDARY OUTCOMES:
SOFA - Sequential Organ Failure Assessment Score up to 15 days after randomization | 15 days
  Sequential Organic Failure Assessment [SOFA]. This will be a primary secondary outcome. Analysis will check for trends in SOFA up to 15 days in a single model.
Need for mechanical ventilation | 30 days (or until hospital discharge)
  Intubation and initiation of mechanical ventilation for any given reason
Duration of mechanical ventilation | 30 days (or until hospital discharge)
  Number of days the patient remains in mechanical ventilation

OTHER OUTCOMES:
Oxygenation index | 14 days
  Daily oxygenation levels assessed using the ROX index [(Oxygen Saturation/Inspired Fraction)/Respiratory Rate] from randomization to discharge or day 14, whichever comes first.
C-reactive protein levels during first 15 days after randomization | 15 days
  C-reactive protein levels over time up to 15 days or hospital discharge.
Lymphocyte/neutrophil ratio during first 15 days after randomization | 15 days
  Lymphocyte/neutrophil ratio over time up to 15 or until discharge discharge day.
D-dimer serum level during first 15 days after randomization | 15 days
  D-dimer serum levels over time or until hospital discharge.
Fibrinogen serum levels during first 15 days after randomization | 15 days
  Fibrinogen serum levels over time up to 15 days or until hospital discharge
Prothrombin Time levels during first 15 days after randomization | 15 days
  Prothrombin Time over time up to 15 days or until hospital discharge.
Activated Partial Thromboplastin Time during first 15 days after randomization | 15 days
  Activated Partial Thromboplastin Time over time up to 15 days or until hospital discharge.
Mortality | 1 year after randomization
  One-year all cause mortality
Euroquol questionnaire for quality of life with 5 dimensions (EQ-5D) | 1 year after randomization
  Quality of Life measured by EQ-5D from 11111-33333, lower values being better

CONTACTS AND LOCATIONS:
Overall Officials: Fernando G Zampieri, MD, Principal Investigator — Research Coordinator; Alexandre B Cavalcanti, Study Chair — Institute Director
Locations (3):
- Brazil (3):
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - BP-A Beneficiência Portuguesa de São Paulo, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data will be available under reasonable request after approval by the steering committee.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol will be available in December, together with analysis plan
Access Criteria: Protocol and analysis plan will be uploaded to Clinicaltrials.gov

REFERENCES:
- [Derived] Zampieri FG, Westphal GA, Santos MAD, Gomes SPC, Gomes JO, Negrelli KL, Santos RHN, Ishihara LM, Miranda TA, Laranjeira LN, Valeis N, Santucci EV, de Souza Dantas VC, Gebara O, Cohn DM, Buchele G, Janiszewski M, de Freitas FG, Dal-Pizzol F, de Matos Soeiro A, Berti IR, Germano A, Schettini DA, Rosa RG, Falavigna M, Veiga VC, Azevedo LCP, Damiani LP, Machado FR, Cavalcanti AB; BRICNet. Antisense therapy to block the Kallikrein-kinin pathway in COVID-19: The ASKCOV randomized controlled trial. J Crit Care. 2024 Dec;84:154892. doi: 10.1016/j.jcrc.2024.154892. Epub 2024 Aug 3. PMID 39096659